CLINICAL TRIAL: NCT02605720
Title: Electrocardiographic Safety Evaluation of Monthly Dihydroartemisinin-Piperaquine for the Use in Mass Treatment Campaigns to Block Malaria Transmission
Brief Title: Cardiac Safety of Repeated Doses of Dihydroartemisinin-Piperaquine for the Use in Mass Treatment Campaigns
Acronym: ECG-Lihir
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Lihir Medical Centre (Other)
Collaborators: Walter and Eliza Hall Institute of Medical Research (Other); Papua New Guinea Institute of Medical Research (Other Government); Barcelona Institute for Global Health (Other)
Responsible Party: Principal Investigator, Oriol Mitja, Assistant Professor, Lihir Medical Centre
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LihirMC
Record Dates: First submitted 2015-11-12; First posted 2015-11-16 (Estimated); Last update posted 2016-03-03 (Estimated); Status verified 2016-02

CONDITIONS: Malaria
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dihydroartemisinin-piperaquine (Experimental)
  Interventions: Drug: Dihydroartemisinin-piperaquine

INTERVENTIONS:
Drug: Dihydroartemisinin-piperaquine — DHA/PPQ dose 2.1/17.1 mg/Kg daily for 3 days (PNG National Malaria Treatment Protocol) monthly for 3 months
  Other Names: Eurartesim

SUMMARY:
Mass drug administration with antimalarial treatment is a tool that can potentially reduce or totally eliminate malaria parasite infections from a population. Dihydroartemisinin-piperaquine (DHA/PPQ) given monthly for 3 months to the entire population might be a good candidate for mass drug administration because the long acting PPQ exerts a long post-treatment prophylactic effect against reinfection and relapse. The use of a repeated dose of DHA/PPQ could lead to increased PPQ plasma concentrations and increased cardiotoxicity. However, there is no data on a second course of treatment or on safety of the drug administered in repeated monthly doses. The proposed project is a clinical trial to assess the electrocardiographic safety of monthly DHA/PPQ (for 3 days at a time) for 3 months. The investigators aim to assess the safety of the drug to be used monthly in mass treatment campaigns. Recommendations issued from this study will benefit health authorities on Lihir-Island by setting the stage for a possible subsequent campaign to completely eliminate malaria from the whole island. This study could be a crucial step to inform the feasibility of drug-based strategies for eliminating malaria elsewhere in PNG, other Melanesian countries and throughout the world.

DETAILED DESCRIPTION:
Given the absence of regulatory data related to the safety of repeated dosing, the European Medicines Agency has set a conservatively long 2-month "wash-out" period before administration of subsequent courses can be recommended. Unfortunately such a recommendation would make it impossible to implement effective mass drug administration with PPQ as this probably requires a maximum interval of one month between doses (in order to ensure that drug levels remain high enough to prevent infections occurring between doses). Therefore it is important that a formal evaluation is performed to regulatory standards that can conclusively document the safety of repeated monthly doses of PPQ. The extensive previous experience from monthly PPQ administration in China suggests that such a study would pose minimal risks to study participants.

Various studies have looked at the potential of DHA/PPQ to cause prolongation of corrected QT interval (QTc) intervals in humans. In a study of 62 adults and children, in Cambodia, electrocardiographic (ECG) findings after DHA/PPQ treatment showed a lengthening of the mean QTc by 11 ms. In two randomized controlled trials in Thailand, the mean QTc prolongation of 56 patients was 14 ms after the last dose of DHA/PPQ. The degree of QT prolongation observed in these studies was therefore similar to that seen with other anti-malarial drugs (including lumefantrine, and chloroquine) generally considered to have no cardiotoxicity in conventional dosing, and substantially less than with others such as halofantrine.and quinidine that have been associated with cardiotoxicity. Study-DM09-006 compared QTc data of healthy subjects that received DHA/PPQ with respective placebo groups and found maximum mean QT Fridericia's correction (QTcF) prolongation of 45.2 ms if co-administered with high fat, and 21.0 ms if fasting (EMEA/H/C/119). Of total of 96 participants given DHA/PPQ in the three studies mentioned above, no subjects showed QTc > 500ms post-treatment or prolongations (after- vs pre-dose) >60ms.

The proposed project is a pharmacovigilance study for electrocardiographic safety evaluation of monthly DHA/PPQ (administered as a conventional 3-day course repeated monthly for 3 months). The investigators aim to assess the safety of the drug to be used monthly in mass treatment campaigns.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female ≥3 years to ≤50 years
2. Good general health by medical history physical examination, baseline electrocardiographs and laboratory tests.
3. No clinically relevant abnormalities in blood pressure and heart rate
4. No clinically relevant abnormalities in 12-lead ECG results*

   *Patients with a QTcB or QTcF greater than 450 ms or clinically significant abnormalities of rhythm at Screening are not eligible. Patients with a pre-dose baseline value > 450 ms should be withdrawn from the study prior to dosing.

   Exclusion Criteria:
5. A history of additional risk factors for Torsades-des-Pointes (e.g., heart failure, hypokalemia, family history of Long QT Syndrome);
6. The use of concomitant medications that prolong the QT/QTc interval;
7. Any condition requiring regular concomitant medication, including herbal products and over-the-counter (OTC) medication or predicted need of any concomitant medication during the study;
8. History of relevant clinical allergic reactions of any origin;
9. Any other condition that in the opinion of the Investigator would interfere with the evaluation of the results or constitute a health risk for the subject;
10. Patients who are not willing to give informed consent (patient and/or parent/legal representative), or who withdraw consent.
11. Pregnant women in the 1st trimester of pregnancy.

Ages: 3 Years to 49 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2015-09; Primary Completion 2016-01 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Change in QTcF interval (Fridericia's correction QT interval) after study drugs administration compared to baseline | Day 58
Plasma piperaquine concentrations after study drugs | Day 58

SECONDARY OUTCOMES:
Change in QTcF interval after study drugs administration compared to baseline | Day 3
Change in QTcF interval after study drugs administration compared to baseline | Day 31

CONTACTS AND LOCATIONS:
Locations (1):
- Lihir medical Centre, Londolovit, New Ireland Province, Papua New Guinea

REFERENCES:
- [Derived] Millat-Martinez P, Salman S, Moore BR, Baro B, Page-Sharp M, Batty KT, Robinson LJ, Pomat W, Karunajeewa H, Laman M, Manning L, Mitja O, Bassat Q. Piperaquine Pharmacokinetic and Pharmacodynamic Profiles in Healthy Volunteers of Papua New Guinea after Administration of Three-Monthly Doses of Dihydroartemisinin-Piperaquine. Antimicrob Agents Chemother. 2022 Aug 16;66(8):e0018522. doi: 10.1128/aac.00185-22. Epub 2022 Jul 6. PMID 35862743